CLINICAL TRIAL: NCT05152914
Title: Intravitreal Enzyme Replacement Therapy to Prevent Retinal Disease Progression in Children With Neuronal Ceroid Lipofuscinosis Type 2 (CLN2)
Brief Title: Intravitreal ERT to Prevent Retinal Disease Progression in Children With CLN2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David L Rogers, MD (Other)
Responsible Party: Sponsor-Investigator, David L Rogers, MD, Chief of the Department of Ophthalmology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001444
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Neuronal Ceroid Lipofuscinosis Type 2
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — cerliponase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Drug: Cerliponase Alfa

INTERVENTIONS:
Drug: Cerliponase Alfa — Brineura is a hydrolytic lysosomal N-terminal tripeptidyl peptidase indicated to slow the loss of ambulation in symptomatic pediatric patients 3 years of age and older with late infantile neuronal ceroid lipofuscinosis type 2 (CLN2), also known as tripeptidyl peptidase 1 (TPP1) deficiency.
  Other Names: Brineura

SUMMARY:
This is a phase I/II randomized, masked, clinical trial to determine the safety and efficacy of intravitreal administration of cerliponase alfa.

DETAILED DESCRIPTION:
This is a Phase I/II study for 5 subjects receiving an intravitreal injection of cerliponase alfa under sedation into the proclaimed study eye(s) in a 4-week interval over 24 months. This study will be monitored by a Data Safety Monitoring Committee (DSMB). Each subject will participate in the ongoing study for an active period of 2 years. Subjects will then transfer to a bi-annual monitoring program where data will be collected from bi-annual standard of care visits for an additional 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Genotypic confirmation of classical CLN2 Batten's disease from a CLIA certified lab.
* Enzyme level deficiency of tripeptidyl-peptidase
* Minimum age requirement: 24 months of age at enrollment
* Maximum age requirement: 72 months of age at enrollment
* Currently receiving intraventricular cerliponase alfa
* Willing to participate in the proposed study visits over the 2-year period
* Minimum central retinal thickness (CRT) of 140μm based upon OCT assessment
* Clear ocular media
* No ocular pathology present to account for vision loss other than optic atrophy and pigmentary retinopathy that is felt to be due to the CLN2 disease process

Exclusion Criteria:

* Any opacities in the clear ocular media including vitreous debris.
* History of ocular trauma or prior ocular surgery.
* Episode of generalized motor status epilepticus within four weeks before the First Dose visit
* Severe infection (e.g., upper respiratory tract infection, pneumonia, pyelonephritis, or meningitis) within four weeks before the First Dose visit (enrollment may be postponed)
* Those with a history of bleeding disorders.
* History of or current chemotherapy, radiotherapy or other immunosuppression therapy within the past 30 days (corticosteroid treatment may be permitted at the discretion of the PI)
* Has a medical condition, or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's wellbeing, safety, or clinical interpretability

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring for the development of unacceptable toxicity. | 2 years
  Based on the development of unacceptable toxicity, defined as the occurrence of any Grade 3 or higher, unanticipated, treatment related toxicity.

SECONDARY OUTCOMES:
Efficacy of intravitreal cerliponase alfa to stabilize fundoscopic features. | 2 years
  Efficacy will be determined by measuring the Weill Cornell LINCL Ophthalmic Severity Score prior to each injection.
Efficacy of intravitreal cerliponase alfa to stabilize retinal architecture. | 2 years
  Efficacy will be determined by measuring central retinal thickness via OCT imaging prior to each injection.

CONTACTS AND LOCATIONS:
Overall Officials: David Rogers, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz A, Kohlschutter A, Mink J, Simonati A, Williams R. NCL diseases - clinical perspectives. Biochim Biophys Acta. 2013 Nov;1832(11):1801-6. doi: 10.1016/j.bbadis.2013.04.008. Epub 2013 Apr 17. PMID 23602993
- [Background] Sleat DE, Donnelly RJ, Lackland H, Liu CG, Sohar I, Pullarkat RK, Lobel P. Association of mutations in a lysosomal protein with classical late-infantile neuronal ceroid lipofuscinosis. Science. 1997 Sep 19;277(5333):1802-5. doi: 10.1126/science.277.5333.1802. PMID 9295267
- [Background] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815
- [Background] Gardner E, Bailey M, Schulz A, Aristorena M, Miller N, Mole SE. Mutation update: Review of TPP1 gene variants associated with neuronal ceroid lipofuscinosis CLN2 disease. Hum Mutat. 2019 Nov;40(11):1924-1938. doi: 10.1002/humu.23860. Epub 2019 Jul 26. PMID 31283065